CLINICAL TRIAL: NCT02559258
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Escalating Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Epsi- Gam in Healthy, Cat-, Dust Mite-, or Bermuda Grass-Allergic Subjects
Brief Title: Escalating Single Dose Study of Epsi- Gam in Healthy Normal Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Tunitas Therapeutics, Inc. (Industry)
Collaborators: Tunitas Therapeutics Australia Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TUN001-101
Record Dates: First submitted 2015-09-02; First posted 2015-09-24 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Allergy and Immunology
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental)
  Interventions: Drug: 0.1 mg/kg epsi-gam or placebo (6:2)
- Cohort 2 (Experimental)
  Interventions: Drug: 0.3 mg/kg epsi-gam or placebo (6:2)
- Cohort 3 (Experimental)
  Interventions: Drug: 1.0 mg/kg epsi-gam or placebo (6:2)
- Cohort 4 (Experimental)
  Interventions: Drug: 3 mg/kg epsi-gam or placebo (6:2)
- Cohort 5 (Experimental)
  Interventions: Drug: 10 mg/kg epsi-gam or placebo (6:2)

INTERVENTIONS:
Drug: 0.1 mg/kg epsi-gam or placebo (6:2) — administered as a single intravenous infusion on Day 1, infused over 30 minutes
  Arms: Cohort 1
Drug: 0.3 mg/kg epsi-gam or placebo (6:2) — administered as a single intravenous infusion on Day 1 infused over 30 minutes
  Arms: Cohort 2
Drug: 1.0 mg/kg epsi-gam or placebo (6:2) — administered as a single intravenous infusion on Day 1 infused over 30 minutes
  Arms: Cohort 3
Drug: 3 mg/kg epsi-gam or placebo (6:2) — administered as a single intravenous infusion on Day 1 infused over 60 minutes
  Arms: Cohort 4
Drug: 10 mg/kg epsi-gam or placebo (6:2) — administered as a single intravenous infusion on Day 1 infused over 120 minutes
  Arms: Cohort 5

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, single-dose, dose- escalation study in otherwise healthy cat-, dust mite-, or Bermuda grass-allergic male and female subjects. There will be five dosing cohorts (0.1, 0.3, 1.0, 3.0 and 10.0 mg/kg), with eight subjects in each cohort, randomized to either epsi-gam (6 subjects) or placebo (2 subjects) for a total of 40 subjects. The first cohort will receive the starting dose of 0.1 mg/kg epsi-gam or placebo and subsequent cohorts will be recruited sequentially to receive escalating doses of epsi-gam or placebo.

ELIGIBILITY:
Eligible subjects must meet all of the following inclusion criteria:

1. Be informed of the nature of the study and provide written informed consent prior to undergoing screening procedures.
2. Be a healthy male of any race or ethnicity, at least 18 years of age and no more than 65 years of age, inclusively, OR
3. Be a healthy female of any race or ethnicity of non-childbearing potential, at least 18 years of age and no more than 65 years of age, inclusively, OR
4. Be a healthy non-pregnant, non-lactating female of any race or ethnicity of childbearing potential, at least 18 years of age and no more than 65 years of age, inclusive, with a negative pregnancy test who agrees to use 2 medically acceptable forms of birth control from Screening through 57 days after receiving study drug.
5. Have a Body Mass Index (BMI) within the range of 18.5 to 30.0 kg/m2.
6. Have a history of allergic reactivity to cats, dust mite, or Bermuda grass as expressed by allergic symptoms including rhinitis.
7. Standardized cat allergenic extract (10,000 BAU/mL, ALK- Abello), dust mite allergenic extract (10,000 AU/mL, ALK- Abello), dust mite allergenic extract (10,000 AU/mL, ALK- Abello), or Bermuda grass allergenic extract (10,000 BAU/mL, ALK- Abello) elicits a wheal at least 5 mm up to approximately 10-15 mm in diameter that exceeds two diluent controls by at least 4 mm.
8. Have allergen-specific IgE for cat, dust mite, or Bermuda grass as measured by ImmunoCAP® with a Class rating of 1 or greater.
9. Histamine reactivity of 3 mm or greater, with surrounding erythema, on testing using a standardized epicutaneous delivery device.
10. Be able and willing to discontinue any first and second generation antihistamine use beginning at least 7 days prior to undergoing initial screening skin puncture tests and throughout study participation.
11. Have baseline spirometry (FEV1, FVC, FEF 25%-75%) with FEV1 ≥ 80% predicted and other values within the normal range.

Exclusion Criteria:

Subjects who meet any of the following criteria must be excluded:

1. Diluent control elicits a wheal ≥ 3 mm on testing.
2. History of severe systemic allergic reactions to cats, dust mite, or Bermuda grass
3. Clinical history of persistent asthma
4. Dermatographism or any skin disorder (i.e., atopic dermatitis) that would make skin testing or proper interpretation impractical.
5. Chronic urticaria.
6. Underlying heart, liver, kidney, or lung disease or any other medical condition such that the subject would be at increased risk for a poor outcome should a generalized allergic or other reaction occur.
7. Any abnormal laboratory value(s) considered to be clinically significant by the Investigator.
8. Use of systemic corticosteroids within the past three months prior to initial screening.
9. Use of topical corticosteroids on the area(s) to undergo skin tests within the past three weeks prior to initial screening.
10. Use of systemic beta-blocking or ACE-inhibiting agents within the past three weeks prior to initial screening.
11. Use of tricyclic antidepressants within the past three weeks prior to initial screening.
12. Use of H2 antagonists within 24 hours prior to initial screening.
13. Use of any agents known or likely to interact with adrenaline.
14. Use of omalizumab (Xolair®) within the past six months prior to enrolment.
15. Pregnant females as determined by a positive serum or urine hCG test.
16. Lactating females.
17. Participation in another experimental drug or device trial and receipt of an investigational product within the past 30 days, five half-lives or twice the duration of the biochemical effect of the investigational product (whichever is longer) prior to dosing in the present study.
18. Any mental impairment as judged by the Investigator that would limit ability to comply with study requirements.
19. History of infection with, or positive screen for, Hepatitis B (HBsAg, Hepatitis B Surface Antigen), Hepatitis C (HCVAb, Hepatitis C Antibody), or Human Immunodeficiency Virus (HIV 1 or 2).
20. Positive urine screen for drugs of abuse. Positive ethanol breath test.
21. Concurrent disease or condition, that, in the opinion of the Investigator, places the subject at high risk of poor treatment compliance or of not completing the study.
22. Has smoked or consumed nicotine-containing products within past 3 months prior to receiving study drug or has a positive urine test for cotinine, and does not agree to refrain from smoking for the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be assessed by monitoring AEs (frequency and severity) and SAEs, vital signs, PFTs | From start of study drug administration through Day 57 (+/- 2 days)
  ECGs, clinical laboratory values (including clinically significant changes from baseline) from blood and urine samples, performing physical examinations and pregnancy tests and reviewing concomitant medications.

CONTACTS AND LOCATIONS:
Locations (1):
- Q-Pharm, Brisbane, Queensland, Australia